CLINICAL TRIAL: NCT02527889
Title: The Effect of Resistive Exercise on Forearm Blood Flow and Tissue Oxygenation Among Breast Cancer Survivors With or at Risk for Breast Cancer-related Lymphoedema (BCRL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Rufina Lau, Clinical Associate, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BCRL-1
Record Dates: First submitted 2015-07-16; First posted 2015-08-19 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Lymphedema; Breast Cancer
Keywords: Exercise; blood flow velocity; tissue oxygenation; BCRL
MeSH Terms: conditions — Lymphedema; Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): The exercise group will receive a supervised resistive exercise training. Subjects in the exercise group will attend small group-based exercise sessions twice a week for 8 weeks supervised by physiotherapists.
  Interventions: Other: Exercise training
- Control Group (No Intervention): The control group will receive no exercise training and continue to receive standard medical care.

INTERVENTIONS:
Other: Exercise training — 8-week resistive exercise training
  Arms: Exercise Group

SUMMARY:
The purpose of the study is to evaluate the effect of resistive exercise on forearm blood flow and tissue oxygenation among breast cancer survivors with or at risk for breast cancer-related lymphoedema (BCRL).

DETAILED DESCRIPTION:
160 subjects who have a diagnosis of breast cancer , 80 with and 80 without BCRL, will be recruited. Eligible subjects are Chinese ethnicity female breast cancer survivors, aged younger than 70 years old and body mass index less than 30kg/m2, remained disease free with a clinical diagnosis of stable BCRL and without BCRL. Subjects will be excluded if they have bilateral or unstable BCRL, defined as significant changes to the arm or receiving intensive therapy (i.e. decongestive therapy or antibiotics for infection) within the past 3 months, or musculoskeletal, cardiovascular and/ or neurological disorders that could inhibit them from exercising.

Primary outcomes include brachial artery blood flow measured by a Doppler ultrasound device and tissue oxygenation measured by near-infrared spectroscopy (NIRS). Additional outcomes and measures include arm circumference measurement, bioelectrical impedance spectroscopy, self-reported lymphoedema symptoms survey, handgrip dynamometer strength testing, upper limb range of motion measurements and quality of life measures using Functional Assessment of Cancer Therapy-Breast Cancer subscale (FACT-B) questionnaire will be obtained.

All outcomes measures will be assessed on both affected and contralateral unaffected arms of all subjects at pre-exercise, immediately post-exercise and 3-month after exercise. Comparison of the baseline measurements between breast cancer survivors with and without BCRL will be obtained.

Subjects will be randomly assigned by computer programme to exercise group and control group. Randomization will be stratified by whether axillary dissection and/ or axilla radiotherapy was given or not. The exercise group will receive supervised resistive exercise programme. Subjects in the exercise group will attend small group-based exercise sessions twice a week for 8 weeks supervised by physiotherapists. The duration of each exercise session will last for approximately 1 hour. Prior to resistive exercises, the subjects will perform warm up with movements of large joints and shoulder girdle for 15 minutes. Resistive exercises will focus on the major muscle groups in the upper body. Loading of resistive exercises will be prescribed and progressed according to individual capacity reaching a level of moderate to high loading (6 -12 repetition maximum). The subjects will also be instructed to perform stretching exercises specific to the muscle groups trained after the session. Symptoms responses will be monitored using self-reported lymphoedema symptoms survey before and after each exercise session. Rate of perceived exertion will also be recorded immediately after each exercise session.

ELIGIBILITY:
Inclusion Criteria:

* female breast cancer survivors
* remained disease free, as defined by unremarkable clinical examination within recent 6 months, with a clinical diagnosis of stable lymphoedema and without lymphedema.

Exclusion Criteria:

* active breast cancer
* have bilateral lymphedema or unstable lymphedema
* have musculoskeletal, cardiovascular and/ or neurological disorders that could inhibit them from exercising.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Brachial artery blood flow | 20 weeks
  Measured by a Doppler ultrasonic device with a linear probe
Tissue oxygenation | 20 weeks
  Measured by Near-infrared spectroscopy

SECONDARY OUTCOMES:
Arm circumference measurement | 20 weeks
  Measured by tape measure at 10cm-interval from the ulnar styloid process
Extent of lymphoedema | 20 weeks
  Measured by bioelectrical impedance spectroscopy
Self-reported lymphoedema symptoms survey | 20 weeks
Hand grip strength | 20 weeks
  Measured by hand grip dynamometer
Upper limb range of motion measurement | 20 weeks
  Measured shoulder range of motion with standard goniometer
Quality of life measures | 20 weeks
  Measured using Functional Assessment of Cancer Therapy - Breast Cancer Subscale (FACT-B) Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong